CLINICAL TRIAL: NCT05410639
Title: Effect of Online Education Given to Parent on Motor Social Development for The Premature Babies in The Neonatal Intensive Care Unites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 09.2020.1352
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2021-12

CONDITIONS: Premature Infant
Keywords: Premature Infant,Motor Development,Social-Communication Development,Parental Stress,Online Education
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Parents of premature infants in the experimental group received online education consist of information to support infants motor,social-communication development.and to manage the parents stress.
  Interventions: Other: online education program
- Control group (Placebo Comparator): The parents of premature babies in the control group did not receive any education programs
  Interventions: Other: no online education program

INTERVENTIONS:
Other: online education program — The training we provided was to give exercises and advice to parents according to the age of the baby in order to stimulate the motor and social development of the baby,and then, an improvement in the stress state of the parents by their participation in the care of their baby.The training, which began with the discharge of the baby from the hospital, was in the form of slide presentations and videos.
  Arms: Study group
Other: no online education program — Parents and their infants in the control group did not receive any online education program
  Arms: Control group

SUMMARY:
Our study aim to evaluate the effect of online program that provides education to parents of premature infants in which stayed in the neonatal intensive care units (NICU),in their motor,socail-communişcation development and the parents stress level.

DETAILED DESCRIPTION:
Our study aim to increase the level f knowledge of the parents of premature infants that stayed in the NICU,to better manage their stress and to provide them with informations to support the motor and social-communication development of their infants.

ELIGIBILITY:
Inclusion Criteria:

* infants Stayed in the neonatal intensive care unit for some time after premature birth for the purpose of care and treatment.
* Being a premature baby born at or under 32 weeks
* infant corrected age between 0-8 months
* To agree to participate in the study.

Exclusion Criteria:

* Having a concomitant major anomaly and genetic disease
* The fact that the family did not accept the evaluation of their baby in motor and social-communication area at sixth month of the study.

Ages: 0 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Alberta Infant Motor Scale (AIMS) | Premature infant motor development was assessed one time by AIMS at their 6 month corrected age
  AIMS assesses the gross infant motor skills in supine, prone, sitting and standing positions with 58 items.the child is scored dec 0 to 58 points and evaluated with age-appropriate percentile curves:0-10 atypical development, 11-25 questionable performance, 26-75 normal performance, 76-90 very good performance, 91-100 are classified as excellent performance.
The Social-Communication Area Screening Test of İnfant (SCASI) | Premature infant social-communication development was assessed one time by SCASI at their 6 month corrected age.
  SCASI assesses the social-communication infant skills,filled by the parents.it is an original and fast test for the early identification and evaluation of children at developmental risk in infancy and early childhood up to the age of 6-24 months.

SECONDARY OUTCOMES:
Parenting Stress Index, Fourth Edition Short Form (PSI-4-SF) | Parents stress level was assessed one time by PSI-4-SF at their infant 6 month corrected age.
  PSI-4-SF assesses the parents stress level.PSI-4-SF contains 36 items: 12 items for Parental Stress (PS) , 12 items for Parent-Child dysfonctional Interaction (P-CDI), and 12 items for Difficult Child (DC).The normal range for scores is within the 16th to 84th percentiles.Scores in the 85th to 89th percentile are considered high,and scores in the 90th percentile or higher are considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Khaoula Ben Kilani, Principal Investigator — Bachelor study principal invistigator Marmara University; Gönül Acar, Study Chair — Assoc.Prof.
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)